CLINICAL TRIAL: NCT01065389
Title: Phase 1 RCT of Progressive Resistance Training on Small Solute Clearance, Functional Capacity and Quality of Life in Intradialysis Patients
Brief Title: Resistance Training in Intradialysis Patients
Acronym: DIAPRE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sikkim Manipal University (Other)
Responsible Party: Principal Investigator, Mr. Baskaran Chandrasekaran, Senior Physiotherapist, Sikkim Manipal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CTRI/2010/091/000014
Record Dates: First submitted 2010-02-04; First posted 2010-02-09 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Dialysis; End Stage Renal Disease
Keywords: Intradialysis; Resistance training; Protein Catabolic Rate; Urea kinetics; Quality of life; VO2 max
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prgressive Resistance Exercise Training (Experimental): Progressive Resistance Exercise Training thrice a week for 12 weeks. For first two weeks, 60% of 5 repetition maximum, progressing at 5% of 5 repetition maximum each week reaching upto 110% of 5 Repetition maximum at the end of 12 weeks
  Interventions: Behavioral: Progressive Resistance Exercise Training
- Unstructured Resistance Exercise (Active Comparator): Unstructured Resistance Exercise thrice a week for 12 weeks. For 12 weeks, 20% 5 repetition maximum (which will not induce training effect and any physiological responses)and free range of motion exercises with no progression.
  Interventions: Behavioral: Unstructured Nonprogressive resistance exercise

INTERVENTIONS:
Behavioral: Progressive Resistance Exercise Training — Progressive Resistance Exercise Training thrice a week for 12 weeks. For first two weeks, 60% of 5 repetition maximum, progressing at 5% of 5 repetition maximum each week reaching upto 110% of 5 Repetition maximum at the end of 12 weeks
  Other Names: Strength Training
  Arms: Prgressive Resistance Exercise Training
Behavioral: Unstructured Nonprogressive resistance exercise — Unstructured Resistance Exercise 30 minutes a day, thrice a week for 12 weeks. For 12 weeks, 20% 5 repetition maximum (which will not induce training effect and any physiological responses)and free range of motion exercises with no progression.
  Other Names: Non progressive strength training
  Arms: Unstructured Resistance Exercise

SUMMARY:
Dialysis patients usually have peripheral muscle weakness due to metabolic disturbances (increased protein catabolism) and fatigue. This muscle weakness may decrease functional capacity and quality of life. It also serves to increase cardiovascular risk factors in these end stage renal disease patients. Peripheral muscle strength training shall combat physical inactivity during dialysis. In the investigators trial, the investigators hypothesis that peripheral muscle training might regulate protein catabolic rate,renal functions, cardiovascular risk factors, improve functional capacity and quality of life in endstage renal disease patients undergoing dialysis.

DETAILED DESCRIPTION:
End stage renal failure patients undergoing dialysis have profound muscle wasting, reduced functional capacity and quality of life due to uremia, steroids, frequent dialysis and fatigue. During dialysis, physical inactivity further deteriorates the patient's functional capacity. Aerobic or strength training may combat this physical inactivity. It may also improve the functional capacity and quality of life. Recent studies have claimed the benefits of resistance exercises in improving functional capacity. But they have not documented effects on kidney function (electrolyte and urea kinetics) and muscle wasting (protein catabolic rate). In our trial, we attempt to study the effects of resistance training in improvement of renal function and muscle wasting apart from functional capacity and quality of life in dialysis patients

ELIGIBILITY:
Inclusion Criteria:

* Must have end stage renal disease (diagnosed and the stage graded by nephrologist or the intensivist concerned) for more than 6 months and dialysis for at least 3 months (the impact of exercise training can be easily assessed)
* Must be between the ages of 30 - 60 years of age/ both genders.
* Must be able to understand the purpose of exercise testing and resistance training.

Exclusion Criteria:

* Those with acute nephritic syndrome and hematuria < 2 months.
* Those with profound anemia and blood transfusion < 2 months
* Those underwent renal transplantation < 6 months.
* Those receiving/ received cytotoxic drugs - amiloride, azathioprine/ aspirin (antiplatelets)< 2 months
* Those with coagulation disorders or under anticoagulants < 4 months.
* Those underwent recent cardiac surgeries and with recent unstable cardiac failures
* Those with recent cerebrovascular accidents < 6 months
* Those have recent urinary tract infections, Renal and bladder carcinomas < 2 months
* Those with absolute contraindications for resistance exercise training (as per American College of Sports Medicine.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-04 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Serum and Urea biochemistry - electrolytes (Na, K+), serum albumin, inflammatory markers, urea kinetics, protein catabolic rate | Bimonthly

SECONDARY OUTCOMES:
Maximal Oxygen Consumption (VO2 max) and Heart Rate Recovery through Queens College step test | Once Monthly
Fat levels by skin fold measurements | Once monthly
Handgrip strength by dynamometer | Once monthly
Six minute walk test distance | Once monthly
Quality of life (KDQOL - SF questionnaire) | Once monthly
Depression (Beck Depression Questionnaire) | Once monthly
Lactate Threshold | Once monthly

CONTACTS AND LOCATIONS:
Overall Officials: Baskaran Chandrasekaran, MPT, Principal Investigator — Lecturer / Consultant cardiopulmonary Physiotherapist; Bidhan C Sharma, MPT, Study Chair — Assistant Professor/ Consultant Physiotherapist; Manish Goon, BPT, Study Chair — Clinical Physiotherapist; Nikita Joshi, MPT, Study Chair — Head of Department/ Associate Professor; Arpan Battacharia, MD, Study Chair — Dialysis Unit Incharge; Bidita Kandelwal, MD, Study Director — Head of Medicine Department
Locations (1):
- Central Referral Hospital, SMIMS, Gangtok, Sikkim, India